CLINICAL TRIAL: NCT04880109
Title: A Phase 2, Double-blind, Placebo-controlled, Efficacy, and Safety Study of APX-115 in Hospitalized Patients With Confirmed Mild to Moderate COVID-19.
Brief Title: A Phase 2 Study of APX-115 in Hospitalized Patients With Confirmed Mild to Moderate COVID-19.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment Challenges
Sponsor: Aptabio Therapeutics, Inc. (Individual)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A01-115-03
Record Dates: First submitted 2021-04-29; First posted 2021-05-10 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: Pulmonary fibrosis; COVID-19; SARS-COV-2; ROS
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis | interventions — isuzinaxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APX-115 (Experimental): Oral administration of APX-115 100mg, daily for 14 days
  Interventions: Drug: APX-115
- Placebo (Placebo Comparator): Oral administration of Placebo, daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APX-115 — Oral administration of APX-115 100 mg capsule once daily for 14 days
  Arms: APX-115
Drug: Placebo — Oral administration of placebo capsule once daily for 14 days
  Arms: Placebo

SUMMARY:
This phase 2 study is to assess the safety and tolerability of APX-115 active doses compared to placebo following multiple oral dosing in hospitalized patients with confirmed, mild to moderate, symptomatic COVID-19. It is anticipated that approximately 80 patients will be randomized into the study in a 1:1 ratio to 100 mg APX-115 or placebo arm.

DETAILED DESCRIPTION:
APX-115 is a potent small molecule inhibitor of NADPH-oxidase (Nox) isozymes being developed by Aptabio Therapeutics Inc. The Nox enzymes represent a family of 7 membrane enzymes (Nox1, Nox2, Nox3, Nox4, Nox5, Duox1, and Duox2) which catalyze NADPH-dependent generation of superoxide and secondary reactive oxygen species (ROS).

ROS are often generated during virus infection, thus promoting apoptosis, lung injury, and inflammation/allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent themselves or through their legally authorized representative.
2. Male or female patients, of any race or ethnicity, 18 to 80 years of age, inclusive, on the day of informed consent. Racial and ethnic minorities should be included in the study population to the greatest extent possible.
3. Laboratory-confirmed SARS-CoV-2 infection as determined within 14 days of randomization by real time RT-PCR or other commercial or public health assay authorized by FDA or other applicable health authority .
4. Onset of COVID-19 symptoms within 14 days prior to randomization.
5. Have at least one of the following symptoms at screening: fever, cough, shortness of breath, myalgia, ageusia, anosmia, fatigue, or weakness.
6. Hospitalized with COVID-19 disease (WHO COVID-19 Clinical Improvement Ordinal Scale score of 3 [hospitalized, no oxygen therapy], 4 [hospitalized, oxygen by mask or nasal prongs], or 5 [high-flow oxygen or non-invasive mechanical ventilation])
7. Patient is aware of the investigational nature of this study and willing to comply with protocol treatments, blood tests, and other evaluations listed in the informed consent form.

Exclusion Criteria:

1. Females who are pregnant (negative pregnancy test required for all women of childbearing potential at screening) or breastfeeding.
2. Male patients and women of childbearing potential (women who are not surgically sterile or postmenopausal defined as postmenopausal for >12 months) who are not using at least one protocol specified method of contraception.
3. COVID-19 disease as defined by the WHO COVID-19 Clinical Improvement Ordinal Scale, scores of 6 (intubation and mechanical ventilation) or 7 (ventilation + additional organ support - pressors, renal replacement therapy, extracorporeal membrane oxygenation).
4. Expected survival less than 72 hours.
5. Treatment with other drugs thought to possibly have activity against SARS CoV 2 infection within 7 days or within 5 half-lives, whichever is longer, prior to enrollment or concurrently. Drugs that have received FDA emergency use authorization or COVID-19 approval are allowed.
6. Treatment with immunosuppressants, combination of 2 or more RAS blockers, UGT inhibitors and inducers, herbal/natural supplements, potassium-sparing diuretic, and radiographic contrast agent prior to enrollment or concurrently.
7. History of abuse of drugs or alcohol that could interfere with adherence to study requirements as judged by the investigator.
8. Use of any other concurrent investigational drugs while participating in the present study.
9. Patient requires frequent or prolonged use of systemic corticosteroids (≥20 mg of prednisone/day or equivalent for >4 weeks) or other immunosuppressive drugs (eg, for organ transplantation or autoimmune conditions).
10. Known renal disease with an estimated glomerular filtration rate <30 mL/min.
11. Patients with clinically apparent liver disease (eg, jaundice, cholestasis, hepatic synthetic impairment, or active hepatitis) or moderate or severe hepatic impairment as determined by Child-Pugh score Class B or C.
12. Alanine aminotransaminase (ALT) or aspartate aminotransaminase (AST) >3 × upper limit of normal (ULN) AND total bilirubin levels >2 × ULN OR ALT or AST >5 × ULN.
13. Total bilirubin >1.5 × ULN, unless the patient has known Gilbert's syndrome.
14. Hemoglobin <9 g/dL for females or <11 g/dL for males.
15. Absolute neutrophil count <1500/mm3.
16. Thrombocytopenia (platelets count <100 × 109/L).
17. Inability to swallow oral medications or a gastrointestinal disorder with diarrhea (eg, Crohn's disease) or malabsorption at screening.
18. Any other clinically significant medical condition or laboratory abnormality that, in the opinion of the investigator, would jeopardize the safety of the patient or potentially impact patient compliance or the safety/efficacy observations in the study.
19. History of an allergic reaction or hypersensitivity to the study drug or any component of the study drug formulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | over the 60-day period
  Adverse events will be assessed to evaluate the safety and tolerability of APX-115 in mild-to-moderate COVID-19 patients. Clinical laboratory evaluations, vital signs, and ECG will be used to assess adverse events.

SECONDARY OUTCOMES:
Time to clinical recovery | Up to 60 Days
  Recovery is defined as when WHO Clinical Improvement Ordinal Scale equal to or less than 3
Time to discharge | Up to Day 60
  WHO Clinical Improvement Ordinal Scale is equal to or less than 2
Time to symptomatic recovery | Up to Day 60
  When none of the COVID-19 Symptom Assessment scores are higher than 1
Time to complete symptomatic recovery | Up to Day 60
  When none of the COVID-19 Symptom Assessment scores are higher than 0
Change in log10 SARS-CoV-2 viral load | Up to Day 14
  hange from baseline in log10 SARS-CoV-2 viral load as measured by RT-PCR by Days 5 and 14
Proportion of patients in clinical recovery | Up to Day 29
  Symptom Assessment
scoring of WHO Clinical Improvement Ordinal Scale | Up to Day 29
  9-point scale on key analysis days for levels ≥3
Changes from baseline in anti-inflammatory markers in blood | Day 1 and Day 14
  Blood will be analyzed for changes from baseline in anti-inflammatory markers, such as C-reactive protein, ferritin, lactate dehydrogenase, D-dimer, troponin, and transforming growth factor-β.
Changes from baseline in pro-inflammatory cytokines in blood | Day 1 and 14
  Blood will be analyzed for changes from baseline in pro-cytokine panel of the blood, such as interleukin (IL)-1β, IL-6, and interferon-γ.
Changes from baseline in 8-isoprostane in blood | Days 1 and 14
  Blood will be analyzed for changes from baseline in 8-isoprostane.
Trough (predose) plasma concentration (Ctrough) | Day 1
  Trough (predose) plasma concentration (Ctrough) will be analyzed from plasma samples for pharmacokinetic assessment of APX-115.
Maximum observed plasma concentration (Cmax) | Days 1, 5, and 14
  Maximum observed plasma concentration (Cmax) will be analyzed from plasma samples for pharmacokinetic assessment of APX-115.
Time to Cmax (Tmax) | Days 1, 5, and 14
  Time to Cmax (Tmax) will be analyzed from plasma samples for pharmacokinetic assessment of APX-115.
Area under the plasma concentration versus time curve (AUC) from time zero to the Time of last quantifiable concentration (AUC0-last) | Days 1, 5, and 14
  Area under the plasma concentration versus time curve (AUC) from time zero to the time of last quantifiable concentration (AUC0-last) will be analyzed from plasma samples for pharmacokinetic assessment of APX-115.
AUC within a dosing interval (AUCtau, where tau = 12 hours) | Days 1, 5, and 14
  AUC within a dosing interval (AUCtau, where tau = 12 hours) will be analyzed from plasma samples for pharmacokinetic assessment of APX-115.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Alternative Research Associates, LLC, Hialeah, Florida
  - Anne Arundel Medical Center, Baltimore, Maryland
  - Millennium Physicians Group, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided